CLINICAL TRIAL: NCT07014943
Title: A Study of High Dose Gemcitabine, Busulfan and Thiotepa With Autologous Stem Cell Transplantation for Primary or Relapse Central Nervous System Lymphomas
Brief Title: High-Dose Gemcitabine, Busulfan, and Thiotepa Followed by ASCT in Primary Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Clinical Professor, Sichuan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GemBuTT-1.0
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)
MeSH Terms: interventions — Gemcitabine; Busulfan; Thiotepa; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine, busulfan and thiotepa as conditioning therapy (Experimental): Gemcitabine (2.5 g/m²) (Days -9 and -3), Busulfan (3.2 mg/kg) (Days -9 to -7), and Thiotepa (5 mg/kg) (Days -5, -4, and -3) were all administered intravenously.
  Interventions: Drug: High dose Gemcitabine, Busulfan, and Thiotepa as conditioning therapy

INTERVENTIONS:
Drug: High dose Gemcitabine, Busulfan, and Thiotepa as conditioning therapy — Gemcitabine (2.5 g/m²) (Days -9 and -3), Busulfan (3.2 mg/kg) (Days -9 to -7), and Thiotepa (5 mg/kg) (Days -5, -4, and -3) were all administered intravenously. Peripheral stem cells were infused on Day 0.

SUMMARY:
The goal of this single-arm, prospective study is to learn if high dose gemcitabine, busulfan and thiotepa with autologous stem cell transplantation to treat primary or relapse central nervous system lymphomas. It will learn about the safety and efficacy of combination therapy. The main question it aims to answer is:

Efficacy and safety of the combination of high dose gemcitabine, busulfan and thiotepa as a bridging therapy to ASCT in patients with CNSL.

Participants will:

Take gemcitabine (2.5 g/m²) was administered intravenously (IV) on Days -9 and -3, Busulfan (3.2 mg/kg) was given IV over 3 hours on Days -9 to -7, and thiotepa (5 mg/kg) was administered IV on Days -5, -4, and -3. Peripheral stem cells were infused on Day 0.

Visit the clinic for checkups and tests in accordance with the International Primary CNS Lymphoma Group (IPCG).

Researchers will observe the patients receiving GemBuTT regimen as conditioning therapy in CNSL.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 70 years;
2. CNS status of complete remission (CR) or partial response (PR) as assessed by magnetic resonance imaging (MRI), positron emission tomography-computed tomography (PET/CT), or CSF analysis (if applicable);
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2;
4. absence of systemic lymphoma in the neck, chest, abdomen, and pelvis as assessed by CT and bone marrow biopsy;
5. negative HIV and hepatitis virus infections (particularly hepatitis B or C, with HBV DNA ≥ 10,000 copies/mL);
6. left ventricular ejection fraction (LVEF) ≥50% and no uncontrolled arrythmias or symptomatic cardiac disease;
7. forced expiratory volume in one second (FEV1) ≥70%;
8. serum creatinine clearance ≥ 50 ml/min and/or serum creatinine ≤ 1.8 mg/dL;
9. serum bilirubin ≤ 2 times the upper limit of normal, serum glutamate oxaloacetate transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) ≤ 3 times the upper limit of normal.

Exclusion Criteria:

1. relapse after stem cell transplantation;
2. other uncontrolled malignancies;
3. immunodeficiency;
4. active infection requiring parenteral antibiotics;
5. pregnant or lactation;
6. severe psychiatric or psychological conditions.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years from ASCT
  The time from stem-cell reinfusion to disease progression, relapse, or death from any cause

SECONDARY OUTCOMES:
OS | 2 years post ASCT
  The time from ASCT to death from any cause
non-relapse mortality (NRM) | 100 days
  NRM was defined as death without evidence of relapse or progression
Hematopoietic recovery | 30 days
  Neutrophil recovery was defined as the first of three consecutive days with an absolute neutrophil count (CAN) ≥ 500/μL (0.5×109/L) after ASCT. Platelet recovery was defined as the first of three consecutive days with a platelet count ≥ 20 000/μL (20 ×109/L) without platelet transfusion for seven consecutive days.
Non-hematological adverse events (AEs) | 2 months
Lymphoma relapse or progression | 2 years
  Relapse or progression was defined as lymphoma progression following ACST

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No